CLINICAL TRIAL: NCT01483768
Title: Evaluation of the Impact of Bariatric Surgery by Sleeve Gastrectomy on Iron Intestinal Absorption in Morbidly Obese Patients
Brief Title: Study of Sleeve Gastrectomy on Iron Intestinal Absorption in Morbidly Obese Patients
Acronym: FORBES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOR 10083
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Iron Deficiency
Keywords: Sleeve gastrectomy; Obesity surgery; Iron deficiency; HEPCIDINE
MeSH Terms: conditions — Obesity; Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A: (Experimental): Sleeve gastrectomy for morbid obesity
  Interventions: Procedure: Sleeve gastrectomy for morbid obesity

INTERVENTIONS:
Procedure: Sleeve gastrectomy for morbid obesity — Sleeve gastrectomy or longitudinal gastrectomy for morbid obesity: is a partial gastrectomy without interruption of the gastric continuity. This procedure includes the resection of the great curvature of the stomach, the fundus , except the lesser curvature and the antrum.
  Other Names: Longitudinal gastrectomy

SUMMARY:
Subject: Evaluation of the impact of obesity surgery by sleeve gastrectomy on intestinal iron absorption of morbid obese subjects.

Control of intestinal absorption of iron is mediated by hepcidin, which is expressed in adipose tissue and that its expression is increased in morbidly obese subjects. The working hypothesis is that this increase could explain the high prevalence of systemic iron depletion observed in obese patients.

Main objective: Assess the impact of the decrease in fat mass induced by surgery in obese patients on the intestinal absorption of iron (evaluated by measuring the expression of iron transporters in the duodenum)

DETAILED DESCRIPTION:
Study Rationale a high prevalence of iron deficiency and anemia has recently been characterized in obese patients and may be related to the stage of low-grade systemic inflammation associated with obesity

Control of intestinal absorption of iron is mediated by hepcidin, a small circulating peptide synthesized primarily by the liver. the synthesis of hepcidin is increased in inflammatory condition and very recently it was shown that hepcidin is expressed in adipose tissue and that its expression is increased in morbidly obese subjects

The working hypothesis is that this increase could explain the high prevalence of systemic iron depletion observed in these patients. the use of bariatric surgery is becoming more common to treat severe obesity (BMI above 35 kg / m2)

The sleeve gastrectomy, recently introduced, involves a very significant weight loss. however, its impact on iron deficiency and anemia are not known

main objective Assess the impact of the decrease in fat mass induced by surgery in obese patients on the intestinal absorption of iron (evaluated by measuring the expression of iron transporters in the duodenum

Secondary objectives:

* Assess the impact of the decrease in fat mass induced by surgery in obese patients on the concentration of circulating hepcidin.
* To study the correlation between the level of expression of iron transporters in the duodenum and the plasma concentration of circulating hepcidin
* Search for a correlation between the level of hepcidin expression in subcutaneous adipose tissue and visceral and concentration of plasma hepcidin before surgery.
* Evaluate the effects of sleeve gastrectomy surgery on haematological and iron status of obese patients.

Selection criteria for patients:

Inclusion criteria: female subjects, having a body mass index > 40 kg/m2 (or > 35 kg/m2 with comorbidity) justifies a obesity surgery, For whom the indication of obesity surgery has been laid, the collective decision is taken in consultation, as part of care between different specialty (physicians, surgeons, psychiatrists ...)

Non-inclusion criteria strictly less than age 18 years or strictly greater than 60 years, history of bariatric surgery or stomach, hepatic cytolysis (transaminases > 3n) during cancer treatment (radio or chemotherapy treatments) coefficient of transferrin saturation > 45%; known history of any of the following: hematologic disease requiring transfusions, hemochromatosis, Wilson's disease (because of known interference between metabolism of iron and copper), Chronic inflammation; Patient did not receive a medical examination; Patient did not give informed consent in writing, not affiliated with Patient Social Security or CMU ( universal health coverage) (recipient or beneficiary), known pregnancy

Number needed: 88 patients enrolled

Total duration of the study: 54 months

Duration of participation for each patient: 24 months

Duration of inclusion: 30 months

Methods:

Prospective open multicenter study cognitive. 4 visits are planned as part of this research with some specificity for the different centers.

Visit 1: Presentation of the study and obtaining consent. Visit 2: consultation with implementation of a multidisciplinary assessment of duodenal biopsies by gastroscopy, additional laboratory tests and a pregnancy test if necessary.

Visit 3: surgery (sleeve gastrectomy) with adipose tissue biopsies. Visit 4: creation of a consultation with multidisciplinary assessment of duodenal biopsies by gastroscopy and additional laboratory tests.

Examinations required specifically for research: duodenal biopsies, additional laboratory tests, biopsies of adipose tissue and pregnancy test (dipstick) for all premenopausal women (contraceptives or not).

Primary assessment criteria:

The intestinal absorption of iron will be assessed by the level of expression of iron transporters (DMT1 and ferroportin) mRNA (messenger ribonucleic acid) level by RT-qPCR (reverse transcription quantification polymerase chain reaction) and at the protein level by Western blot.

secondary assessment (s) criteria (s) The concentration of hepcidin plasma will be measured by ELISA in adipose tissue, the level of hepcidin expression is quantified by RT-qPCR .

The haematological will assess the presence of anemia (hemoglobin less than 12g/dl) its micro or macrocytic hemolytic and / or regenerative

ELIGIBILITY:
Inclusion Criteria:

* morbid obese women selected for bariatric surgery

Exclusion Criteria:

* non obese patients, less than 18 years old, haematological disease with need of blood transfusions

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2012-09-25 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The intestinal absorption of iron | Time Frame 1 year (Time point(s) at which outcome measure is assessed):
  The intestinal absorption of iron will be assessed by the level of expression of iron transporters (DMT1 and ferroportin) mRNA level by RT-qPCR and at the protein level by Western blot.

CONTACTS AND LOCATIONS:
Overall Officials: Simon MSIKA, MD, Ph D, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Colombes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided